CLINICAL TRIAL: NCT03725397
Title: Inpatient Versus Outpatient Foley Cervical Ripening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000022710
Record Dates: First submitted 2018-06-22; First posted 2018-10-31 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Induced; Birth
MeSH Terms: interventions — Inosine Monophosphate

STUDY DESIGN:
Intervention Model Description: two cohort double blinded clinical trial
Who Masked: Participant
Masking Description: randomized double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatients with a transcervical Foley catheter (Experimental): Women with a transcervical Foley catheter in place that will spend the night at home.
  Interventions: Behavioral: Outpatient
- Inpatients with a transcervical Foley catheter (Active Comparator): Women to be admitted to the hospital overnight which has been a "standard of care".
  Interventions: Behavioral: Inpatient

INTERVENTIONS:
Behavioral: Outpatient — The offered (studied) intervention will be allowing the women with a transcervical Foley catheter in place to spend the night at home.
  Arms: Outpatients with a transcervical Foley catheter
Behavioral: Inpatient — Women with a transcervical Foley catheter to be admitted to the hospital overnight which has been a "standard of care".
  Arms: Inpatients with a transcervical Foley catheter

SUMMARY:
To compare the efficacy and safety of cervical ripening with transcervical Foley catheter in inpatient vs outpatient setting

DETAILED DESCRIPTION:
The aim of the current study is to compare the efficacy and safety of cervical ripening with transcervical Foley catheter in inpatient vs outpatient setting in a diverse, urban population within the United States. We hypothesize that there will be no differences in time-to-delivery, failed induction rates, cesarean section rates, or maternal/neonatal morbidity and that there will be no differences in total length of stay (LOS), hours of sleep, active labor duration, and perceived satisfaction between groups.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Induction of Labor is present
* Gestational age > 37 completed weeks with absence of comorbidities with an optimal dating (ultrasonography was performed before 22 weeks gestation)
* Singleton fetus in cephalic presentation confirmed with an ultrasound at the time of presentation for induction of labor
* Cervical exam with Bishop Score <6
* Intact membranes
* Normal vital signs (blood pressure < 140/90, normal body temperature) at the time of presentation for Induction of Labor and within the last 24 hours
* Maternal age ≥18 years of age

Exclusion Criteria:

* Any contraindication for vaginal birth by institutional policy
* Multiple gestation
* History of cesarean delivery
* Oligohydramnios/polyhydramnios/anhydramnios (MVP <2cm)
* Rupture of membranes
* Poorly controlled diabetes (Hgb A1C>8% and/or fingerstick glucose above target >50% of the time in the past week)
* Poorly controlled chronic hypertension, gestational hypertension or preeclampsia (patient requiring IV antihypertensives within 4 hours of arrival)
* Vaginal bleeding
* Any conditions that require continuous electronic fetal monitoring either by institutional policy or provider determination (intrahepatic cholestasis of pregnancy, intrauterine growth restriction, abnormal non-stress test, others)
* Fetal anomaly with anticipated neonatal intensive care unit admission
* Fetal demise
* HIV infection, presence of genital herpetic lesion
* History of substance abuse during this pregnancy
* History of precipitous delivery (delivery <3hrs from onset of labor)
* Poor access to care (social, distance to hospital > 45 min, limited transportation)
* Poor social situation, history of domestic violence, untreated/uncontrolled psychiatric condition
* Inability to give informed consent, history of mental retardation
* Strong preference for inpatient management
* Inability to understand English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women of diverse ethnic and social background who are at term and have medical indications for delivery and who are recommended to undergo cervical ripening followed by induction of labor. These will be women who are generally healthy and their pregnancy has been uncomplicated.
Enrollment: 54 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Time of Foley catheter extrusion | within 24 hours
  Antepartum time of Foley catheter extrusion before patient being brought to labor

SECONDARY OUTCOMES:
Bishop score | during labor
  Bishop scoring system used to consider having cervical ripening.Women with favorable cervices (BS 8 or more) are considered to have a cervix ripe and ready to proceed to induction. BS <6 are considered unripe, and therefore may benefit from additional ripening modalities
Total time in cervical ripening | from labor induction to delivery time
  Measure of total time in cervical ripening
Total time slept during pre-induction | during labor
  Total time slept during pre-induction
Total time in hospital | no max but an average of 3 days
  Total time in hospital
Analgesia used during pre-induction | within 24 hours before Pitocin initiation
  Analgesia used during pre-induction
Use of oxytocin | 3 days
  Pitocin is given as a continuous infusion and the dose is titrated according to the contraction pattern (goal max contractions but not hyperstimulation). We will calculate the total time of Pitocin infusion as well as total dose (rate of infusion x time).
Fever over 38 degrees C | within 7 days of Foley placement
  Did the patient have a fever over 38 degrees C
Neonatal Intensive Care Unit (NICU) | within 7 days of Foley placement
  Was the baby admitted to NICU
APGAR scores | 1 minute of life
  Apgar score is a universal (international) scoring system. The 1-minute score determines how well the baby tolerated the birthing process. The 5-minute score tells the health care provider how well the baby is doing outside the mother's womb.
APGAR scores | 5 minutes of life
  Apgar score is a universal (international) scoring system. The 1-minute score determines how well the baby tolerated the birthing process. The 5-minute score tells the health care provider how well the baby is doing outside the mother's womb.
Hospital charges | within 30 days after discharge
  All patients will be charged. We are hoping to see lower charges for women in the Out Patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kohari, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital- St. Raphael, New Haven, Connecticut
  - Yale New Haven Hospital, York Street Campus, New Haven, Connecticut

REFERENCES:
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803